CLINICAL TRIAL: NCT02405143
Title: Electrical Stimulation for Restoration of Vision After Stroke in the Damaged Visual Field of Patients With Unilateral Stroke (REVIS Helsinki)
Brief Title: Restoration of Vision After Stroke
Acronym: REVIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Academy of Finland (Other)
Responsible Party: Principal Investigator, Turgut Tatlisumak, MD, PhD, FAHA, FESO, Associate Professor, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UAK1010001
Record Dates: First submitted 2015-02-06; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Stroke; Infarction; Posterior Cerebral Artery; Hemianopsia
Keywords: Controlled clinical trial; Electric Stimulation Therapy
MeSH Terms: conditions — Stroke; Infarction, Posterior Cerebral Artery; Hemianopsia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active tACS using DC-Stimulator MC (Experimental): 15 to 30 patients will be randomized to the arm receiving the active transcranial alternating current stimulation (tACS) treatment using DC-Stimulator MC.
  Interventions: Device: Active tACS using DC-Stimulator MC
- Sham stimulation using DC-Stimulator MC (Sham Comparator): The same number of patients as in the active arm, 15 to 30, will be randomized to receive sham stimulation using DC-Stimulator MC.
  Interventions: Device: Sham stimulation using DC-Stimulator MC

INTERVENTIONS:
Device: Active tACS using DC-Stimulator MC — Transcranial alternating current stimulation (tACS) is administered using DC-Stimulator MC (NeuroConn GmbH, Ilmenau Germany). Stimulation is administered through two 5 cm2 saline-soaked electrodes placed in the Fpz position and on the right arm. Stimulation will consist of short blocks, during which stimulation frequency will be ramped up to 30Hz with maximum current of 1.5mA. Stimulation will be administered for 20 minutes on 10 consecutive weekdays.
  Arms: Active tACS using DC-Stimulator MC
Device: Sham stimulation using DC-Stimulator MC — Patients in the sham group will undergo the same preparations as the treatment group. This includes using an identical electrode placement and session duration as for the experimental arm. In order to create the effect of phosphenes, one 5Hz current burst per minute will be administered using the individual phosphene threshold of the patient. This is not expected to have therapeutic effects.
  Arms: Sham stimulation using DC-Stimulator MC

SUMMARY:
Occipital stroke is associated with homonymous visual field defects (occurring on one side of the visual field). Despite spontaneous recovery, some degree of defect is often permanent. Currently, no treatment exists for such visual field defects.The purpose of this study is to test the efficacy of a type of electrical brain stimulation method, transcranial alternating current stimulation, in reducing these type of visual field defects in their chronic stage.

ELIGIBILITY:
Inclusion Criteria:

* Occipital ischemic or hemorrhagic stroke 6 months or older
* Hemianopia or quadrantanopia demonstrated by standard automated perimetry
* Visual field defect is stable across baseline
* Presence of residual vision and detectable gradual transition between the the intact and absolutely blind parts of the visual field
* Best corrected visual acuity for at least one eye better or equal to 0.4

Exclusion Criteria:

* Eye or central nervous system disease that interferes with the study
* Cardiac pacemaker
* Other metallic devices or implants precluding participation in MRI scans
* Pregnancy or lactation period
* Epileptic seizures in the past 10 years
* Use of antiepileptic or sedative drugs
* Expected low compliance due to substance abuse
* Known active malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Improved detection in the visual field defined as the percentage change of the stimulus detection rate in High-resolution perimetry (HRP) | Change between 3-7 days pre-treatment, at 3-7 days post-treatment, and at 2 months post-treatment
  HRP is a computer-based perimetry using a supra-threshold stimulus. It is used to detect residual vision between the absolute defect and seeing field and to monitor subtle changes in perceptual ability. HRP is performed in fixation control using an eye tracker.
  The primary outcome measure will be the percentage change in HRP detection accuracy between pre-test and post-test measurements.

SECONDARY OUTCOMES:
The change in extent of visual fields in standard automated perimetry | Change between 3-7 days pre-treatment, at 3-7 days post-treatment, and at 2 months post-treatment
  A secondary outcome measure will be the change in extent of visual fields i.e. mean threshold measured by means of standard automated perimetry.

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Tatlisumak, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Central Hospital, Helsinki, Finland